CLINICAL TRIAL: NCT02175771
Title: A 26-Week Open-Label Study to Assess the Long-Term Safety of Fluticasone Propionate Multidose Dry Powder Inhaler and Fluticasone Propionate/Salmeterol Multidose Dry Powder Inhaler in Patients 12 Years of Age and Older With Persistent Asthma
Brief Title: Long-Term Safety Study of Fluticasone Propionate (Fp) Multidose Dry Powder Inhaler (MDPI) and Fluticasone Propionate/Salmeterol (FS) MDPI in Patients With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSS-AS-305
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Persistent Asthma
MeSH Terms: interventions — Fluticasone; Salmeterol Xinafoate; Fluticasone-Salmeterol Drug Combination; Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (8):
- Fp MDPI 100 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 200 mcg Fp for 26 weeks. This was the mid-strength experimental intervention in the inhaled corticosteroid (ICS) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol HFA
- FLOVENT HFA 110 mcg (Active Comparator): Participants took 2 inhalations using a hydrofluoroalkane (HFA) inhaler twice a day of fluticasone propionate (Fp) for a total daily dose of 440 mcg Fp for 26 weeks. This was the mid-strength active comparator intervention in the inhaled corticosteroid (ICS) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FLOVENT HFA; Drug: albuterol/salbutamol HFA
- Fp MDPI 200 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate (Fp) for a total daily dose of 400 mcg Fp for 26 weeks. This was the high-strength experimental intervention in the inhaled corticosteroid (ICS) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: Fp MDPI; Drug: albuterol/salbutamol HFA
- FLOVENT HFA 220 mcg (Active Comparator): Participants took 2 inhalations using a hydrofluoroalkane (HFA) inhaler twice a day of fluticasone propionate (Fp) for a total daily dose of 880 mcg Fp for 26 weeks. This was the high-strength active comparator intervention in the inhaled corticosteroid (ICS) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FLOVENT HFA; Drug: albuterol/salbutamol HFA
- FS MDPI 100/12.5 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate/salmeterol (FS) 100/12.5 mcg for a total daily dose of 200/25 mcg FS for 26 weeks. This was the mid-strength experimental intervention in the inhaled corticosteroid/long-acting beta2-agonist (ICS/LABA) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FS MDPI; Drug: albuterol/salbutamol HFA
- ADVAIR DISKUS 250/50 mcg (Active Comparator): Participants took 1 inhalation of a dry-powder formulation twice a day of fluticasone propionate/salmeterol (FS) 250/50 mcg for a total daily dose of 500/100 mcg FS for 26 weeks. This was the mid-strength active comparator intervention in the inhaled corticosteroid/long-acting beta2-agonist (ICS/LABA) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: ADVAIR DISKUS; Drug: albuterol/salbutamol HFA
- FS MDPI 200/12.5 mcg (Experimental): Participants took 1 inhalation using a multidose dry powder inhaler (MDPI) twice a day of fluticasone propionate/salmeterol (FS) 200/12.5 mcg for a total daily dose of 400/25 mcg FS for 26 weeks. This was the high-strength experimental intervention in the inhaled corticosteroid/long-acting beta2-agonist (ICS/LABA) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: FS MDPI; Drug: albuterol/salbutamol HFA
- ADVAIR DISKUS 500/50 mcg (Active Comparator): Participants took 1 inhalation of a dry-powder formulation twice a day of fluticasone propionate/salmeterol (FS) 500/50 mcg for a total daily dose of 1000/100 mcg FS for 26 weeks. This was the high-strength active comparator intervention in the inhaled corticosteroid/long-acting beta2-agonist (ICS/LABA) cohort.
  Albuterol/salbutamol HFA metered dose inhaler (MDI) was supplied to participants throughout the study to be used as needed as a rescue medication.
  Interventions: Drug: ADVAIR DISKUS; Drug: albuterol/salbutamol HFA

INTERVENTIONS:
Drug: Fp MDPI — Fp MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate dispersed in a lactose monohydrate excipient.
  During the treatment period, participants were randomized to either 100 mcg or 200 mcg of Fp one inhalation twice a day for a total daily dose of 200 mcg or 400 mcg. Study drug was administered in the morning and in the evening.
  Other Names: fluticasone propionate; inhaled corticosteroid
  Arms: Fp MDPI 100 mcg; Fp MDPI 200 mcg
Drug: FS MDPI — FS MDPI is an inhalation-driven multidose dry powder inhaler (MDPI) containing fluticasone propionate (Fp) and salmeterol xinafoate (Sx) dispersed in a lactose monohydrate excipient.
  During the treatment period, participants were randomized to either Fp/Sx MDPI 100/12.5 mcg or Fp/Sx MDPI 100/12.5 mcg twice a day for a total daily dose of 200/25 mcg or 400/25 mcg Fp/Sx. Study drug was administered in the morning and in the evening.
  Other Names: fluticasone propionate; inhaled corticosteroid; Salmeterol xinafoate; β2 adrenoceptor agonist
  Arms: FS MDPI 100/12.5 mcg; FS MDPI 200/12.5 mcg
Drug: FLOVENT HFA — FLOVENT HFA is a hydrofluoroalkane (HFA) inhaler containing fluticasone propionate.
  During the treatment period, participants were randomized to either 110 mcg or 220 mcg of FLOVENT two puffs, twice a day for a total daily dose of 440 mcg or 880 mcg. Study drug was administered in the morning and in the evening.
  Other Names: fluticasone propionate; inhaled corticosteroid
  Arms: FLOVENT HFA 110 mcg; FLOVENT HFA 220 mcg
Drug: ADVAIR DISKUS — ADVAIR DISKUS contains a dry powder formulation of fluticasone propionate (Fp) and salmeterol xinafoate (Sx) in a lactose excipient.
  During the treatment period, participants were randomized to Fp 250 mcg/Sx 50 mcg or Fp 500 mcg/Sx 50 mcg one inhalation, twice a day for a total daily dose of 500/100 mcg or 1000/100 mcg. Study drug was administered in the morning and in the evening.
  Other Names: fluticasone propionate; inhaled corticosteroid; salmeterol xinafoate; β2 adrenoceptor agonist
  Arms: ADVAIR DISKUS 250/50 mcg; ADVAIR DISKUS 500/50 mcg
Drug: albuterol/salbutamol HFA — A short-acting β2-adrenergic agonists (SABA), albuterol/salbutamol hydrofluoroalkane (HFA) metered dose inhaler (MDI), was provided to be used as needed for the relief of asthma symptoms during both the run-in and treatment periods (to replace the subject's current rescue medication).
  Other Names: ProAir HFA; short-acting β2-adrenergic agonists

SUMMARY:
The primary objective of the study is to evaluate the long-term safety of fluticasone propionate (Fp) inhalation powder in 2 strengths and fluticasone propionate/salmeterol inhalation (FS) powder in 2 strengths when administered with the Teva multidose dry powder inhaler (MDPI) device over 26 weeks in patients with persistent asthma.

DETAILED DESCRIPTION:
This was a stratified, randomized, open-label, active drug-controlled Phase 3 study.

Patients who met all of the inclusion criteria and none of the exclusion criteria at the screening visit completed a 14 day (±2 days) pretreatment run in period. During the run-in period, patients continued using their current asthma medications (ie, inhaled corticosteroid and/or other controller therapies) except for their SABA, which was replaced by the sponsor-provided albuterol (salbutamol) hydrofluoroalkane (HFA) inhaler to be used as needed for symptomatic relief of asthma symptoms during the run in and treatment periods.

Patients were assigned to inhaled corticosteroid (ICS) monotherapy or inhaled corticosteroid/long acting beta2 agonist (ICS/LABA) combination therapy and then to a mid- or high-treatment strength based on their current asthma maintenance therapy regimen. Patients in each strength of the ICS monotherapy cohort were randomly assigned in a 3:1 distribution to either the Fp MDPI or FLOVENT HFA treatment arm. Patients in each strength of the ICS/LABA combination cohort were randomly assigned in a 3:1 distribution to either the FS MDPI or ADVAIR DISKUS treatment arm. There was a total of 8 treatment arms following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Best pre-bronchodilator forced expiratory volume in 1 second (FEV1) of greater than 40% of their predicted normal value.
2. Patients must have a treatment regimen that includes a short-acting β2 agonist (SABA) (albuterol) for use as needed and either an inhaled corticosteroid (ICS) or an ICS/long-acting β2 agonist (LABA) as a preventative treatment for a minimum of 8 weeks before the SV. Patients currently taking low-dose ICS without LABA are not eligible for this study. Patients currently taking low-dose ICS/LABA may only be entered into the mid ICS strength. All patients must have been maintained on a stable dose of ICS or ICS/LABA for 4 weeks prior to the SV (or pre-SV if necessary) at 1 qualifying doses
3. To meet reversibility of disease criteria, the patient must demonstrate a ≥12% reversibility of FEV1 (and 200 mL for patients aged18 years and older) within 30 minutes following 4 inhalations of albuterol at the SV. Historic reversibility within the past 12 months of the SV may be used to meet this criterion.
4. Written informed consent/assent is obtained. For adult patients (aged 18 years and older, or as applicable per local regulations), the written informed consent form (ICF) must be signed and dated by the patient before conducting any study-related procedure. For minor patients (aged 12 to 17 years, or as applicable per local regulations), the written ICF must be signed and dated by the parent/legal guardian and the written assent form must be signed and dated by the patient (if applicable) before conducting any study-related procedure. Note: Age requirements are as specified by local regulations.
5. Outpatient >= 12 years of age on the date of consent/assent. .
6. Asthma diagnosis: The patient has a diagnosis of asthma as defined by the National Institutes of Health (NIH). The asthma diagnosis has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in medication) for at least 30 days before providing informed consent.
7. The patient is able to perform acceptable and repeatable spirometry.
8. The patient is able to perform peak expiratory flow (PEF) with a handheld peak flow meter.
9. The patient is able to use a metered-dose inhaler (MDI) device without a spacer device and a MDPI device.
10. The patient is able to withhold (as judged by the investigator) his or her regimen of ICS or study drug, and rescue medication for at least 6 hours before the SV and before all treatment visits where spirometry is performed.
11. The patient/parent/legal guardian/caregiver is capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements.
12. SABAs: All patients must be able to replace their current SABA with albuterol/salbutamol HFA inhalation aerosol at the SV for use as needed for the duration of the study.
13. Female patients may not be pregnant, breastfeeding, or attempting to become pregnant.

    * -Other criteria may apply, please contact the investigator for more information

Exclusion Criteria:

1. The patient has a history of a life-threatening asthma exacerbation that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnea, respiratory arrest, or hypoxic seizures.
2. The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the study.
3. The patient has participated as a randomized patient in any investigational drug study within the 30 days preceding the SV (or prescreening visit, as applicable) or plans to participate in another investigational drug study at any time during this study.
4. The patient has previously participated in an Fp MDPI or FS MDPI study.
5. The patient has a known hypersensitivity to any corticosteroid, salmeterol, or any of the excipients in the study drug or rescue medication formulation (ie, lactose).
6. The patient has been treated with any known strong cytochrome P450 (CYP) 3A4 inhibitors (eg, azole antifungals, ritonavir, or clarithromycin) within 30 days before the SV or plans to be treated with any strong CYP3A4 inhibitor during the study.
7. The patient has been treated with any of the prohibited medications during the prescribed (per protocol) washout periods before the SV.
8. The patient currently smokes or has a smoking history of 10 pack-years or more (a pack-year is defined as smoking 1 pack of cigarettes/day for 1 year). The patient may not have used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco).
9. The patient has a culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that has not resolved at least 2 weeks before the SV.
10. The patient has a history of alcohol or drug abuse within 2 years preceding the SV.
11. The patient has had an asthma exacerbation requiring systemic corticosteroids within 30 days before the SV, or has had any hospitalization for asthma within 2 months before the SV.
12. Initiation or dose escalation of immunotherapy (administered by any route) is planned during the study period. However, patients who initiated immunotherapy 90 days or more before the SV and have been on a stable (maintenance) dose for 30 days or more before the SV may be considered for inclusion.
13. The patient has used immunosuppressive medications within 4 weeks before the SV.
14. The patient is unable to tolerate or unwilling to comply with the appropriate washout periods and withholding of all applicable medications. (Patients that require continuous treatment with β-blockers, monoamine oxidase inhibitors, tricyclic antidepressants, anticholinergics, and/or systemic corticosteroids are excluded).
15. The patient has untreated oral candidiasis at the SV. Patients with clinical visual evidence of oral candidiasis who agree to receive treatment and comply with appropriate medical monitoring may enter the study.
16. The patient has a history of a positive test for human immunodeficiency virus, active hepatitis B virus, or hepatitis C infection.
17. The patient is either an employee or an immediate relative of an employee of the clinical investigational center.
18. A member of the patient's household is participating in the study at the same time. However, after the enrolled patient completes or discontinues participation in the study, another patient from the same household may be screened.
19. The patient has a disease/condition that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.

    * Other criteria may apply, please contact the investigator for more information

Criteria for Randomization:

Patients were randomized into the study if they met all of the following criteria:

1. The patient continued to be in general good health, meeting the entry criteria.
2. The patient continued to have a predose/pre-albuterol FEV1 at the randomization visit (RV) that was ≥40% of predicted normal.
3. The patient had no clinically significant abnormal laboratory test results or ECG findings at the screening visit.
4. The patient had no significant changes in asthma medications during run-in, excluding the albuterol/salbutamol HFA (90 mcg ex actuator) or equivalent used as rescue medication as supplied per protocol.
5. The patient did not have a upper respiratory tract infection (URI) or lower respiratory tract infection (LRI) during the run in period. Patients who developed a URI or LRI during the run in period could be discontinued from the study and allowed to re-screen 2 weeks after resolution of symptoms.
6. The patient had no asthma exacerbation during the run in period, defined as any worsening of asthma requiring any significant treatment other than rescue albuterol/salbutamol HFA (90 mcg ex actuator) or equivalent or the patient's run-in MDPI. This included requiring the use of systemic corticosteroids and/or emergency department (ED) visit or hospitalization or an increase in the patient's regularly prescribed nonsteroidal maintenance treatment. Urgent care/ED visits where the treatment was limited to a single dose of nebulized albuterol/salbutamol did not meet the criteria of an asthma exacerbation.
7. The patient had no clinical visual evidence (on oropharyngeal examination) of oropharyngeal candidiasis.
8. The patient did not experience an adverse event that would result in failure to continue to meet selection criteria.
9. The patient did not use any of the prohibited concomitant medications during the run in period.
10. The patient complied with completion of the daily diary, defined as follows:

    * completion of AM and PM asthma symptom scores on 4 or more of the 7 days immediately preceding the RV.
    * completion of rescue medication use (whether used or not) on 4 or more of the 7 days immediately preceding the RV.
    * completion of AM peak expiratory flow (PEF) measurements on 4 or more of the 7 days immediately preceding the RV.
    * recording of AM and PM asthma inhalation therapy use on 4 or more of the 7 days immediately preceding the RV.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 758 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (101):
- United States (101):
  - Teva Investigational Site 12068, Birmingham, Alabama
  - Teva Investigational Site 12112, Mobile, Alabama
  - Teva Investigational Site 12130, Pell City, Alabama
  - Teva Investigational Site 12119, Little Rock, Alaska
  - Teva Investigational Site 12076, Phoenix, Arizona
  - Teva Investigational Site 12135, Scottsdale, Arizona
  - Teva Investigational Site 12132, Tucson, Arizona
  - Teva Investigational Site 12102, Fountain Valley, California
  - Teva Investigational Site 12104, Fresno, California
  - Teva Investigational Site 12123, Fullerton, California
  - Teva Investigational Site 12103, Huntington Beach, California
  - Teva Investigational Site 12073, Long Beach, California
  - Teva Investigational Site 12077, Mission Viejo, California
  - Teva Investigational Site 12098, Napa, California
  - Teva Investigational Site 12149, Northridge, California
  - Teva Investigational Site 12081, Orange, California
  - Teva Investigational Site 12100, Rancho Mirage, California
  - Teva Investigational Site 12133, Riverside, California
  - Teva Investigational Site 12146, Riverside, California
  - Teva Investigational Site 12075, Rolling Hills Estates, California
  - Teva Investigational Site 12074, San Diego, California
  - Teva Investigational Site 12150, San Diego, California
  - Teva Investigational Site 12064, San Jose, California
  - Teva Investigational Site 12061, Stockton, California
  - Teva Investigational Site 12141, Walnut Creek, California
  - Teva Investigational Site 12043, Denver, Colorado
  - Teva Investigational Site 12051, Denver, Colorado
  - Teva Investigational Site 12091, Waterbury, Connecticut
  - Teva Investigational Site 12078, Fort Lauderdale, Florida
  - Teva Investigational Site 12140, Hialeah, Florida
  - Teva Investigational Site 12066, Kissimmee, Florida
  - Teva Investigational Site 12120, Miami, Florida
  - Teva Investigational Site 12127, Miami, Florida
  - Teva Investigational Site 12148, Miami, Florida
  - Teva Investigational Site 12114, Ocala, Florida
  - Teva Investigational Site 12055, Sarasota, Florida
  - Teva Investigational Site 12048, Tallahassee, Florida
  - Teva Investigational Site 12122, Tamarac, Florida
  - Teva Investigational Site 12086, Winter Park, Florida
  - Teva Investigational Site 12111, Gainesville, Georgia
  - Teva Investigational Site 12070, Lawrenceville, Georgia
  - Teva Investigational Site 12072, Marietta, Georgia
  - Teva Investigational Site 12106, Coeur d'Alene, Idaho
  - Teva Investigational Site 12117, Eagle, Idaho
  - Teva Investigational Site 12065, River Forest, Illinois
  - Teva Investigational Site 12059, Shiloh, Illinois
  - Teva Investigational Site 12056, Overland Park, Kansas
  - Teva Investigational Site 12138, Fort Mitchell, Kentucky
  - Teva Investigational Site 12092, Owensboro, Kentucky
  - Teva Investigational Site 12087, Covington, Louisiana
  - Teva Investigational Site 12095, Bangor, Maine
  - Teva Investigational Site 12042, Baltimore, Maryland
  - Teva Investigational Site 12124, Baltimore, Maryland
  - Teva Investigational Site 12052, North Dartmouth, Massachusetts
  - Teva Investigational Site 12139, Minneapolis, Minnesota
  - Teva Investigational Site 12137, Plymouth, Minnesota
  - Teva Investigational Site 12079, Columbia, Missouri
  - Teva Investigational Site 12067, Rolla, Missouri
  - Teva Investigational Site 12057, St Louis, Missouri
  - Teva Investigational Site 12060, St Louis, Missouri
  - Teva Investigational Site 12108, St Louis, Missouri
  - Teva Investigational Site 12128, Warrensburg, Missouri
  - Teva Investigational Site 12136, Bellevue, Nebraska
  - Teva Investigational Site 12115, Las Vegas, Nevada
  - Teva Investigational Site 12131, Las Vegas, Nevada
  - Teva Investigational Site 12126, Ocean City, New Jersey
  - Teva Investigational Site 12129, Verona, New Jersey
  - Teva Investigational Site 12058, Rochester, New York
  - Teva Investigational Site 12113, Rockville Centre, New York
  - Teva Investigational Site 12047, Charlotte, North Carolina
  - Teva Investigational Site 12085, Charlotte, North Carolina
  - Teva Investigational Site 12144, Winston-Salem, North Carolina
  - Teva Investigational Site 12053, Canton, Ohio
  - Teva Investigational Site 12094, Cincinnati, Ohio
  - Teva Investigational Site 12105, Cincinnati, Ohio
  - Teva Investigational Site 12107, Sylvania, Ohio
  - Teva Investigational Site 12069, Tiffin, Ohio
  - Teva Investigational Site 12045, Oklahoma City, Oklahoma
  - Teva Investigational Site 12080, Oklahoma City, Oklahoma
  - Teva Investigational Site 12083, Oklahoma City, Oklahoma
  - Teva Investigational Site 12062, Eugene, Oregon
  - Teva Investigational Site 12097, Medford, Oregon
  - Teva Investigational Site 12049, Portland, Oregon
  - Teva Investigational Site 12134, Bryn Mawr, Pennsylvania
  - Teva Investigational Site 12090, Philadelphia, Pennsylvania
  - Teva Investigational Site 12089, Providence, Rhode Island
  - Teva Investigational Site 12088, Warwick, Rhode Island
  - Teva Investigational Site 12096, Charleston, South Carolina
  - Teva Investigational Site 12147, Spartanburg, South Carolina
  - Teva Investigational Site 12121, Dallas, Texas
  - Teva Investigational Site 12099, El Paso, Texas
  - Teva Investigational Site 12071, Live Oak, Texas
  - Teva Investigational Site 12054, San Antonio, Texas
  - Teva Investigational Site 12145, Waco, Texas
  - Teva Investigational Site 12046, Murray, Utah
  - Teva Investigational Site 12041, South Burlington, Vermont
  - Teva Investigational Site 12125, Richmond, Virginia
  - Teva Investigational Site 12101, Seattle, Washington
  - Teva Investigational Site 12109, Spokane, Washington
  - Teva Investigational Site 12044, Tacoma, Washington
  - Teva Investigational Site 12082, Greenfield, Wisconsin

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Mansfield L, Yiu G, Sakov A, Liu S, Caracta C. A 6-month safety and efficacy study of fluticasone propionate and fluticasone propionate/salmeterol multidose dry powder inhalers in persistent asthma. Allergy Asthma Proc. 2017 Jul 24;38(4):264-276. doi: 10.2500/aap.2017.38.4061. Epub 2017 May 24. PMID 28540844
- [Derived] Miller DS, Yiu G, Hellriegel ET, Steinfeld J. Dose-ranging study of salmeterol using a novel fluticasone propionate/salmeterol multidose dry powder inhaler in patients with persistent asthma. Allergy Asthma Proc. 2016 Jul;37(4):291-301. doi: 10.2500/aap.2016.37.3963. Epub 2016 May 27. PMID 27216137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 1087 patients screened, 758 patients at 103 investigational centers in the US met entry criteria. 331 patients were not enrolled: 267 due to inclusion/exclusion criteria, 21 withdrew consent, 9 were lost to follow up, 4 had an adverse event, and 30 patients had reason of 'other' or missing.
Pre-assignment Details: Participants in each strength of the ICS monotherapy cohort were randomly assigned in a 3:1 distribution to either the Fp MDPI or FLOVENT HFA treatment arm. Participants in each strength of the ICS/LABA combination cohort were randomly assigned in a 3:1 distribution to either the FS MDPI or ADVAIR DISKUS treatment arm.
Groups:
- Enrolled Patients: During the run-in period, patients continued using their current asthma medications (ie, inhaled corticosteroid and/or other controller therapies) except for their short acting beta2-agonist (SABA), which was replaced by the sponsor-provided study rescue medication.
Period: Run-In Period (Pre-assignment)
Arm/Group | Enrolled Patients | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Started | 758 (Enrolled; two participants were enrolled but had no enrollment date in their records.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 674 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 84 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomization criteria not met | 23 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Exclusion criteria met | 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion criteria not met | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Enrolled Patients | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Started | 0 | 127 | 42 | 126 | 41 | 120 | 41 | 133 | 44
Completed | 0 | 111 | 35 | 113 | 36 | 110 | 36 | 116 | 38
Not Completed | 0 | 16 | 7 | 13 | 5 | 10 | 5 | 17 | 6
Not completed — Adverse Event | 0 | 2 | 1 | 1 | 1 | 3 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 9 | 3 | 6 | 2 | 4 | 2 | 9 | 2
Not completed — Noncompliance | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Disease progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Other | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety population which included all randomized participants who received at least 1 dose of randomized study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg | Total
Number analyzed (Participants) | 127 | 42 | 126 | 41 | 120 | 41 | 133 | 44 | 674
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 19 | 7 | 16 | 3 | 13 | 5 | 9 | 1 | 73
  Adults (18-64 years) | 96 | 32 | 96 | 35 | 94 | 31 | 106 | 41 | 531
  Adults (65+ years) | 12 | 3 | 12 | 3 | 13 | 5 | 18 | 2 | 68
  Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 49 | 16 | 46 | 16 | 36 | 21 | 61 | 21 | 266
  Female | 78 | 26 | 78 | 25 | 84 | 20 | 72 | 23 | 406
  Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 118 | 39 | 100 | 33 | 99 | 36 | 112 | 39 | 576
  Hispanic or Latino | 9 | 3 | 24 | 8 | 21 | 5 | 20 | 5 | 95
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 110 | 26 | 99 | 36 | 99 | 32 | 95 | 31 | 528
  Black or African American | 16 | 13 | 22 | 5 | 19 | 9 | 31 | 12 | 127
  Asian | 1 | 1 | 1 | 0 | 2 | 0 | 4 | 0 | 9
  American Indian or Alaskan Native | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  Pacific Islander | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3
  Other | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Missing | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
History of Smoking [Count of Participants; unit: Participants]
  Prior smoker | 26 | 10 | 20 | 5 | 23 | 7 | 24 | 8 | 123
  No tobacco use | 101 | 32 | 106 | 36 | 97 | 34 | 109 | 36 | 551

OUTCOME MEASURES:

1. Primary Outcome: Participants With Treatment-Emergent Adverse Experiences (TEAE) During the Treatment Period
Description: An adverse event was defined as any untoward medical occurrence that develops or worsens in severity during the conduct of a clinical study and does not necessarily have a causal relationship to the study drug. Severity was rated by the investigator on a scale of mild, moderate and severe, with severe= an AE which prevents normal daily activities. Relationship of AE to treatment was determined by the investigator. Serious AEs include death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, OR an important medical event that jeopardized the patient and required medical intervention to prevent the previously listed serious outcomes.
Time Frame: Day 1 to Week 26 of the Treatment Period
Population: Safety population which included all randomized participants who received at least 1 dose of randomized study drug.
  The randomization allocation ratio of 3:1 (study drug: active comparator) should be taken into account when comparing treatment groups within treatment/strength cohorts
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 127 | 42 | 125 | 41 | 120 | 41 | 133 | 44
Participants
  >=1 TEAE | 85 | 29 | 83 | 29 | 92 | 29 | 86 | 30
  >=1 severe TEAE | 8 | 3 | 11 | 3 | 8 | 1 | 12 | 3
  >=1 treatment-related TEAE | 10 | 2 | 6 | 5 | 9 | 4 | 11 | 8
  >=1 severe treatment-related TEAE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=1 serious TEAE | 7 | 2 | 8 | 3 | 6 | 2 | 13 | 3
  >=1 TEAE leading to withdrawal | 2 | 1 | 0 | 1 | 3 | 2 | 0 | 1
  >=1 nonserious TEAE | 85 | 27 | 82 | 29 | 91 | 28 | 85 | 29
  >=1 TEAE resulting in death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Participants With Positive Swab Test Results for Oral Candidiasis
Description: Oropharyngeal examinations for visual evidence of oral candidiasis were conducted at each visit by a qualified healthcare professional. Any visual evidence of oral candidiasis during the oropharyngeal exam was evaluated by obtaining and analyzing a swab of the suspect area.
  This outcomes indicates how many participants had positive swab test results. The total number of participants who had oropharyngeal exams at each timepoint are specified in the timepoint field. Appropriate therapy was to be initiated immediately at the discretion of the investigator and was not to be delayed for culture confirmation. Participants with a culture-positive infection could continue participation in the study on appropriate anti-infective therapy, provided this therapy was not prohibited by the protocol.
Time Frame: Baseline (Day 1 pre-treatment), Weeks 2, 6, 10, 14, 18, 22 26, Endpoint
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 127 | 42 | 125 | 41 | 120 | 41 | 133 | 44
Participants
  Baseline (n=127, 42, 124, 41, 120, 41, 133, 44) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2 (n=123, 42, 123, 40, 117, 39, 131, 43) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 2
  Week 6 (n=119, 41, 119, 40, 115, 39, 125, 43) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0
  Week 10 (n=119, 37, 118, 39, 115, 39, 120, 40) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
  Week 14 (n=116, 36, 115, 38, 113, 38, 120, 41) | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 1
  Week 18 (n=111, 37, 115, 38, 109, 38, 117, 40) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Week 22 (n=110, 36, 113, 36, 110, 37, 116, 38) | 1 | 0 | 1 | 1 | 1 | 0 | 2 | 2
  Week 26 (n=111, 35, 113, 36, 110, 36, 116, 38) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0
  Endpoint (n=125, 42, 123, 41, 119, 40, 132, 44) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0

3. Secondary Outcome: Participants With Potentially Clinically Significant Abnormal Vital Signs During the Treatment Period
Description: Data represents participants with potentially clinically significant (PCS) vital sign values during the Treatment period.
  Significance criteria:
  * Systolic blood pressure - high: >=180 and increase >=20 mmHg
  * Systolic blood pressure - low: <=90 and decrease >=20 mmHg
  * Diastolic blood pressure - high: >=105 and increase of >=15 mmHg
  * Diastolic blood pressure - low: <=50 and decrease of >=15 mmHg
  * Pulse - high: >=120 and increase of >= 15 beats/minute from baseline
  * Pulse - low: <=50 and decrease of >=15 beats/minute
Time Frame: Baseline (Day 1 pre-treatment), Weeks 2, 6, 10, 14, 18, 22 26, Endpoint
Population: Safety population of participants with a baseline and postbaseline vital sign value.
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 125 | 42 | 123 | 41 | 119 | 40 | 132 | 44
Participants
  >=1 abnormality | 5 | 0 | 0 | 1 | 2 | 0 | 2 | 0
  Systolic blood pressure - high | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Systolic blood pressure - low | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Diastolic blood pressure - high | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Diastolic blood pressure - low | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Pulse - high | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse - low | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Shifts From Baseline to Endpoint in Electrocardiogram (ECG) Findings
Description: A 12 lead ECG was conducted at the screening visit and week 26 or the early termination visit. A qualified physician at a central diagnostic center was responsible for interpreting the ECG. The worst post-baseline finding for the participant is summarized. Endpoint refers to the last observation carried forward.
Time Frame: Screening (Day -14), Endpoint (week 26 if study was completed)
Population: Safety population of participants with both screening and endpoint ECGs
Measure: Count of Participants; unit: Participants
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 112 | 39 | 116 | 39 | 116 | 38 | 125 | 39
Participants
  Baseline normal - Endpoint normal | 89 | 31 | 93 | 33 | 90 | 30 | 101 | 28
  Baseline normal - Endpoint abnormal | 8 | 5 | 6 | 1 | 9 | 2 | 8 | 3
  Baseline abnormal - Endpoint normal | 4 | 1 | 4 | 2 | 12 | 2 | 9 | 4
  Baseline abnormal - Endpoint abnormal | 11 | 2 | 13 | 3 | 5 | 4 | 7 | 4

5. Secondary Outcome: Analysis of 24-Hour Urine Cortisol Free Over the 26-Week Treatment Period
Description: Samples for 24-hour urine cortisol were collected at baseline (Day 1, pretreatment), and Weeks 14 and 26. For participants requiring early termination (ET), this evaluation was performed at the ET visit. For participants requiring ET for safety reasons, the visit was not delayed in order to collect the 24-hour urine cortisol.
  The analysis is based on a mixed model for repeated measures (MMRM) model with adjustment for visit, treatment, and a treatment*visit interaction. The urine cortisol result is log transformed prior to analysis and the results are back transformed after modeling. An unstructured covariance matrix is used in the MMRM model.
Time Frame: Baseline (Day 1, pre-treatment), Weeks 14 and 26 and early termination visit if applicable
Population: A urine cortisol analysis subset of the safety population was defined that included participants whose urine samples did not have confounding factors at any visit that could affect the interpretation of the results.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/24 hours
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 80 | 28 | 93 | 28 | 87 | 29 | 91 | 38
mcg/24 hours | 18.45 [15.77 to 21.58] | 13.94 [10.67 to 18.22] | 14.14 [12.23 to 16.34] | 17.50 [13.40 to 22.85] | 17.56 [15.13 to 20.38] | 18.29 [14.07 to 23.77] | 13.02 [11.23 to 15.09] | 15.42 [12.27 to 19.38]
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs FLOVENT HFA 110 mcg; Mid-strength comparison; Test type: Superiority; geometric mean ratio = 1.32, 90% CI 2-sided [1.02 to 1.72] — Fp MDPI / FLOVENT HFA
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs FLOVENT HFA 220 mcg; High-strength comparison; Test type: Superiority; geometric mean ratio = 0.81, 90% CI 2-sided [0.63 to 1.04] — Fp MDPI / FLOVENT HFA
Statistical Analysis 3: Comparison: FS MDPI 100/12.5 mcg vs ADVAIR DISKUS 250/50 mcg; Mid-strength comparison; Test type: Superiority; geometric mean ratio = 0.96, 90% CI 2-sided [0.75 to 1.24] — FS MDPI / ADVAIR DISKUS
Statistical Analysis 4: Comparison: FS MDPI 200/12.5 mcg vs ADVAIR DISKUS 500/50 mcg; High-strength comparison; Test type: Superiority; geometric mean ratio = 0.84, 90% CI 2-sided [0.67 to 1.06] — FS MDPI / ADVAIR DISKUS

6. Secondary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Minute (FEV1) Over the 26-Week Treatment Period
Description: Spirometry measurements were obtained before the AM dose of study drug for the randomization visit (Day 1), at each of the treatment visits and at the early termination visit if applicable. At each visit where FEV1 was assessed, the highest acceptable results from each session were recorded.
  The analysis is based on a mixed model for repeated measures (MMRM) with adjustment for baseline FEV1, sex, age, (pooled) investigational center, visit, treatment, and treatment-by-visit. An unstructured covariance matrix is used in the MMRM model.
Time Frame: Baseline (Day 1 pre-treatment), Weeks 2, 6, 10, 14, 18, 22 26, early termination visit if applicable
Population: The full analysis set (FAS) included all participants in the intent-to-treat (ITT) population who received at least 1 dose of study drug and had at least 1 post-baseline trough FEV1 assessment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Fp MDPI 100 mcg | FLOVENT HFA 110 mcg | Fp MDPI 200 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | ADVAIR DISKUS 250/50 mcg | FS MDPI 200/12.5 mcg | ADVAIR DISKUS 500/50 mcg
Number analyzed (Participants) | 123 | 42 | 120 | 41 | 119 | 40 | 130 | 44
liters | 0.062 (0.0243) | 0.053 (0.0415) | 0.077 (0.0246) | 0.090 (0.0415) | 0.116 (0.0251) | 0.117 (0.0419) | 0.100 (0.0235) | 0.041 (0.0399)
Statistical Analysis 1: Comparison: Fp MDPI 100 mcg vs FLOVENT HFA 110 mcg; Mid-strength comparison; Test type: Non-Inferiority — The study had reasonable power for demonstrating non-inferiority of the study drug to the comparator drug within each cohort. The statistical analysis plan specified that non-inferiority would be demonstrated if the lower limit of the 2-sided 95% confidence interval (CI) for the treatment difference was greater than -125 mL; p = 0.8451, mixed model for repeated measures; LSM difference = 0.009, 95% CI 2-sided [-0.084 to 0.103], Standard Error of Mean 0.0476 — Fp MDPI / FLOVENT HFA
Statistical Analysis 2: Comparison: Fp MDPI 200 mcg vs FLOVENT HFA 220 mcg; High-strength comparison; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.7877, mixed model for repeated measures; LSM difference = -0.013, 95% CI 2-sided [-0.107 to 0.081], Standard Error of Mean 0.0479 — Fp MDPI / FLOVENT HFA
Statistical Analysis 3: Comparison: FS MDPI 100/12.5 mcg vs ADVAIR DISKUS 250/50 mcg; Mid-strength comparison; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.9966, mixed model for repeated measures; LSM difference = 0.000, 95% CI 2-sided [-0.095 to 0.095], Standard Error of Mean 0.0485 — FS MDPI / ADVAIR DISKUS
Statistical Analysis 4: Comparison: FS MDPI 200/12.5 mcg vs ADVAIR DISKUS 500/50 mcg; High-strength comparison; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; p = 0.2056, mixed model for repeated measures; LSM difference = 0.059, 95% CI 2-sided [-0.032 to 0.150], Standard Error of Mean 0.0464 — FS MDPI / ADVAIR DISKUS

ADVERSE EVENTS:
Time Frame: Day 1 to Week 26
Arm/Group | ADVAIR DISKUS 250/50 mcg | ADVAIR DISKUS 500/50 mcg | FLOVENT HFA 110 mcg | FLOVENT HFA 220 mcg | FS MDPI 100/12.5 mcg | FS MDPI 200/12.5 mcg | Fp MDPI 100 mcg | Fp MDPI 200 mcg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/44 | 0/42 | 0/41 | 0/120 | 0/133 | 0/127 | 0/125
Serious Adverse Events (participants affected / at risk) | 2/41 | 3/44 | 2/42 | 3/41 | 6/120 | 13/133 | 7/127 | 8/125
Other Adverse Events (participants affected / at risk) | 22/41 | 23/44 | 24/42 | 25/41 | 70/120 | 68/133 | 65/127 | 55/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADVAIR DISKUS 250/50 mcg (N=41) | ADVAIR DISKUS 500/50 mcg (N=44) | FLOVENT HFA 110 mcg (N=42) | FLOVENT HFA 220 mcg (N=41) | FS MDPI 100/12.5 mcg (N=120) | FS MDPI 200/12.5 mcg (N=133) | Fp MDPI 100 mcg (N=127) | Fp MDPI 200 mcg (N=125)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (4) | 8 (9) | 6 (6) | 4 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADVAIR DISKUS 250/50 mcg (N=41) | ADVAIR DISKUS 500/50 mcg (N=44) | FLOVENT HFA 110 mcg (N=42) | FLOVENT HFA 220 mcg (N=41) | FS MDPI 100/12.5 mcg (N=120) | FS MDPI 200/12.5 mcg (N=133) | Fp MDPI 100 mcg (N=127) | Fp MDPI 200 mcg (N=125)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (4) | 3 (3) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 4 (4) | 6 (7) | 5 (7) | 5 (5)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 5 (6) | 7 (7) | 3 (3) | 10 (10) | 8 (8)
Nasopharyngitis (Infections and infestations) | 4 (5) | 4 (6) | 7 (8) | 5 (6) | 15 (21) | 12 (13) | 17 (20) | 13 (19)
Oral candidiasis (Infections and infestations) | 2 (3) | 5 (9) | 0 (0) | 5 (5) | 5 (8) | 5 (5) | 6 (8) | 5 (5)
Sinusitis (Infections and infestations) | 4 (4) | 8 (9) | 3 (5) | 3 (3) | 9 (12) | 14 (15) | 15 (16) | 6 (7)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 6 (8) | 12 (13) | 8 (10) | 21 (27) | 24 (26) | 23 (36) | 17 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (15) | 2 (4) | 2 (2) | 1 (2) | 9 (11) | 3 (3) | 5 (5) | 6 (13)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (6) | 14 (17) | 8 (13) | 10 (10) | 13 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6) | 5 (6) | 1 (1) | 7 (8) | 9 (9) | 13 (14) | 6 (7)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (2) | 1 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 7 (8) | 2 (3) | 1 (1) | 2 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.